CLINICAL TRIAL: NCT01564004
Title: Clinical Hypnosis Versus Neuro-linguistic Programming Before External Cephalic Version (ECV) - a Prospective Off-centre Randomised Controlled Trial
Brief Title: Clinical Hypnosis Before External Cephalic Version (ECV)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, PD Dr. med. Joscha Reinhard, MBBS BSc(Hon), Principle Investigator, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12/11
Record Dates: First submitted 2012-03-24; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Breech Presentation at Term
Keywords: breech presentation at term; pregnancy; external cephalic version (ECV); clinical hypnosis; neuro-linguistic programming (NLP)
MeSH Terms: interventions — Hypnosis; Neurolinguistic Programming

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical hypnosis (Experimental): 20 minutes tape recorded clinical hypnosis intervention
  Interventions: Other: Clinical hypnosis or neuro-linguistic programming
- Neuro-linguistic programming (Active Comparator): 20 minutes tape recording of nouro-linguistic programming intervention
  Interventions: Other: Clinical hypnosis or neuro-linguistic programming

INTERVENTIONS:
Other: Clinical hypnosis or neuro-linguistic programming — 20 minutes tape recording intervention

SUMMARY:
Does clinical hypnosis or neuro-linguistic programming improve the success rate of external cephalic version?

DETAILED DESCRIPTION:
Prospective off-center randomisation of clinical hypnosis or neuro-linguistic programming intervention prior to a external cephalic version treatment.

ELIGIBILITY:
Inclusion Criteria:

* singleton
* breech presentation
* gestation age above 36 weeks + 6 days

Exclusion Criteria:

* multiples
* cannot understand German language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Successful ECV | 3 hours after ECV treatment
  Rate of cephalic presentation three hours after external cephalic version.

SECONDARY OUTCOMES:
Questionnaire | before and 30 minutes after ECV

CONTACTS AND LOCATIONS:
Locations (1):
- Department of obstetrics and gynaecology, Johann Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany